CLINICAL TRIAL: NCT06501118
Title: Optimizing Care in Critically Ill at UCHealth by Liberalizing the Target O2 in Mechanically-ventilated ICU Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24-0065
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Failure; Acute Hypoxemic Respiratory Failure; Acute Hypoxic Respiratory Failure; Hypoxemia; Hypoxia; Hypoxic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency; Hypoxia | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational intervention (Other): SP02 target ranges will be 90-96%. Education about the specific oxygen targets will be provided to the clinical teams. Real time feedback on adherence to the Sp02 target range will be provided by virtual respiratory therapists.
  Interventions: Other: Education
- Educational intervention Epic alert (Other): An education-based intervention that also focuses on mitigating Occult Hypoxemia in mechanically ventilated patients, and thus utilizes the same patient population. The second intervention will notify the clinical team to an abnormal laboratory result in real time. This laboratory result is already located in the patient's Epic chart under arterial blood gas (ABG), arterial oxygen saturation (Sa02) Patient level randomization will occur in Epic as
  1. alert (notification) the providers of sustained occult hypoxemia or
  2. silent alert The investigators are observing physician behavior in response to alerting them that a patient has occult hypoxemia via an Epic alert.
  Interventions: Behavioral: Epic notification alert

INTERVENTIONS:
Other: Education — 1) Standardized materials to discuss the rationale and procedural aspects of the intervention, including details on the specific oxygen target-related modifications to the mechanical ventilation order-set prior to starting the intervention phase.
  Arms: Educational intervention
Behavioral: Epic notification alert — An education-based intervention that focuses on mitigating Occult Hypoxemia in mechanically ventilated patients and thus utilizes the same patient population. The second intervention will notify the clinical team to an abnormal laboratory result in real time. This laboratory result is already located in the patient's Epic chart under arterial blood gas (ABG), arterial oxygen saturation (Sa02) Patient level randomization will occur in Epic to as
  1. alert (notification) the providers of sustained occult hypoxemia
  2. silent alert
  Arms: Educational intervention Epic alert

SUMMARY:
A multimodal educational intervention to target an oxygen saturation target range (SpO2 90-96%) will reduce ventilator length of stay and reduce occult hypoxemia by increased awareness and adherence to a designated oxygen saturation target range.

DETAILED DESCRIPTION:
This project will be a multi-hospital, cluster randomized study to implement a targeted oxygen saturation (SpO2) range of 90-96% in adult patients receiving mechanical ventilation (MV) using a multimodal educational intervention strategy. Hospital-level randomization to receive the intervention will occur sequentially for a phased roll-out of multimodal education and real-time informatics tools to enhance adherence of the targeted SpO2 range in eligible mechanically ventilated patients. This phased roll-out is achieved through a stepped wedge approach in a one-way crossover design in which all participating hospital ICUs will ultimately implement the intervention, and the timing of the intervention implementation is randomly ordered. The intervention will occur using 4 clusters that switch from control to intervention at 4 pre-determined time points, 1 for each cluster. For each switch, the design incorporates a 2-week transition period for staff education/implementation at each cluster, during which training will be delivered to each participating hospital to improve implementation. The investigators will provide standardized education and materials to local stakeholders for hospital and ICU-level implementation. During the transition period, the cluster cannot be considered as either receiving the structured usual care intervention (education-based intervention) or the unstructured usual care control (current state, no education-based intervention), and thus patients treated in the hospital during that period will not be enrolled or included in the analysis.

The investigators define a targeted SpO2 range (90-96%), PaO2 (60-100 mmHg) target based on thresholds defined in recent published work that incorporates expert opinions from the field and includes consensus among critical care COGG members that represent UCHealth hospitals throughout the North, South, and Metro regions as well as the site locations at which the intervention is proposed to occur. The oxygen target range will be defined by an oxygen saturation (SpO2) 90-96%, and when arterial blood gases are available, an arterial oxygen pressure (PaO2) 60-100 mmHg. The intervention will start when patients requiring mechanical ventilation arrive to an ICU in a participating hospital and the intervention will continue for any period of invasive mechanical ventilation required during ICU stay. A project goal is to achieve adherence to >95% of eligible patient-hours spent in the target SpO2 range, excluding time on FiO2 30% when above SpO2 96% or time on FiO2 100% when below SpO2 90%. Each hospital site will contribute pre-implementation (control) and post-implementation (intervention) data, with the start of the consensus-based intervention period defined by the randomized timing in the stepped wedge design.

Patients will be ventilated with a standardized UCHealth-wide mechanical ventilation order-set to achieve these SpO2 and PaO2 goals. These order-sets included the ARDSNetwork low- and high-PEEP/FiO2 arms, as well as developed protocols for alternative modes of ventilation, such as APRV which can be used at the provider teams' discretion.

Once all hospital clusters have transitioned to the intervention phase, a nested study will commence that involves a patient-level intervention for mechanically ventilated patients experiencing residual occult hypoxemia among participating UCHealth ICUs. These patients will be identified automatically in the EHR (EPIC) by comparing the SaO2 from an ABG laboratory procedure to contemporaneous SpO2 flowsheet row values and then will be randomized 1:1 to either an active or silent notification delivered in real-time to members of the provider team alerting them to each OH instance, with a 12-hour notification lockout. A unique research study order will be created in EPIC for this nested study to facilitate tracking of outcomes for patients randomized to silent and active notification arms in coordination with a health data compass analyst (HDC).

Educational interventions will include:

1. Standardized materials to discuss the rationale and procedural aspects of the intervention, including details on the specific oxygen target-related modifications to the mechanical ventilation order-set prior to starting the intervention phase.
2. EPIC-generated push notification to (1) alert providers in real-time to the presence of OH in their patient with a time-stamp based on SpO2 and SaO2 values compared from vital signs and arterial blood gas oxygen saturation respectively, and (2) inform them of the potential associations of OH with worse outcomes in similar, critically ill patients, and (3) choices for potential changes to management, including an "acknowledge only" option

ELIGIBILITY:
Inclusion Criteria:

* Admission to ICU and requiring invasive mechanical ventilation

Exclusion Criteria:

* Transferred patients from outside the UCHealth system*:
* Patients with pre-existing disease that requires chronic use of positive pressure ventilation delivered through a tracheostomy*:
* Pregnant women:
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3600 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Ventilator Free Days | 30 Days
  The number of days the patient will be free of mechanical ventilation

SECONDARY OUTCOMES:
instances of occult hypoxemia | 30 days
  arterial oxygen saturation below 88% when the Sp02 is 92-96% within 10 minutes identified among all patients
ICU free days | 90 days
  Number of days patients are not in the ICU
Hospital free days | 90 DAYS
  number of days patients are not hospitalized
90 Day in hospital mortality | 90 days
  Patients that die in the hospital before day 90
Time to Mortality to day 90 | 90 Days
  Patients that die within 90 days
Oxygen status at discharge | 90 days
  What if any oxygen the patient is on at discharge
Incidence of needing high level 02 support | 90 days
  The number of times that the patients is in need of heated-high flow nasal cannula (HHFNC) / non-invasive positive pressure ventilation (NIPPV)) after extubation
Discharge disposition | 90 days
  Place the patient is discharged to
Changes to mechanical ventilation order set | 4 hours
  Quantify the number of changes made to the ventilator order set to attempt to deliver more oxygen to the blood. This will capture FIO2, PEEP, Tidal Volume, Inspiratory Pressure changes as a summary numerical unit of measure.
Medication changes | 4 hours
  Addition or dose change of a medication to try and eliminate occult hypoxemia will be quantified numerically. The investigators will include diuretics, inhaled vasodilators, corticosteroids, Intravenous sedatives, and intravenous paralytics in this summary statistic.
Additional procedures in response to occult hypoxemia | 4 hours
  The investigators will quantify the number of additional procedures that may be performed in response to occult hypoxemia. Chest X-ray, Chest CT Scan, arterial blood gas, and placement of arterial catheter procedures will be included in this summary statistic.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Aggarwal, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dylla L, Douin DJ, Anderson EL, Rice JD, Jackson CL, Bebarta VS, Lindsell CJ, Cheng AC, Schauer SG, Ginde AA. A multicenter cluster randomized, stepped wedge implementation trial for targeted normoxia in critically ill trauma patients: study protocol and statistical analysis plan for the Strategy to Avoid Excessive Oxygen (SAVE-O2) trial. Trials. 2021 Nov 8;22(1):784. doi: 10.1186/s13063-021-05688-6. PMID 34749762
- [Background] Semler MW, Casey JD, Lloyd BD, Hastings PG, Hays MA, Stollings JL, Buell KG, Brems JH, Qian ET, Seitz KP, Wang L, Lindsell CJ, Freundlich RE, Wanderer JP, Han JH, Bernard GR, Self WH, Rice TW; PILOT Investigators and the Pragmatic Critical Care Research Group. Oxygen-Saturation Targets for Critically Ill Adults Receiving Mechanical Ventilation. N Engl J Med. 2022 Nov 10;387(19):1759-1769. doi: 10.1056/NEJMoa2208415. Epub 2022 Oct 24. PMID 36278971
- [Background] Racial Bias in Pulse Oximetry Measurement. N Engl J Med. 2021 Dec 23;385(26):2496. doi: 10.1056/NEJMx210003. No abstract available. PMID 34936755
- [Background] Douin DJ, Anderson EL, Dylla L, Rice JD, Jackson CL, Wright FL, Bebarta VS, Schauer SG, Ginde AA. Association Between Hyperoxia, Supplemental Oxygen, and Mortality in Critically Injured Patients. Crit Care Explor. 2021 May 14;3(5):e0418. doi: 10.1097/CCE.0000000000000418. eCollection 2021 May. PMID 34036272
- [Background] Hussey MA, Hughes JP. Design and analysis of stepped wedge cluster randomized trials. Contemp Clin Trials. 2007 Feb;28(2):182-91. doi: 10.1016/j.cct.2006.05.007. Epub 2006 Jul 7. PMID 16829207
- [Background] Panwar R, Capellier G, Schmutz N, Davies A, Cooper DJ, Bailey M, Baguley D, Pilcher V, Bellomo R. Current oxygenation practice in ventilated patients-an observational cohort study. Anaesth Intensive Care. 2013 Jul;41(4):505-14. doi: 10.1177/0310057X1304100412. PMID 23808511
- [Background] Rachmale S, Li G, Wilson G, Malinchoc M, Gajic O. Practice of excessive F(IO(2)) and effect on pulmonary outcomes in mechanically ventilated patients with acute lung injury. Respir Care. 2012 Nov;57(11):1887-93. doi: 10.4187/respcare.01696. Epub 2012 May 15. PMID 22613692
- [Background] Suzuki S, Eastwood GM, Peck L, Glassford NJ, Bellomo R. Current oxygen management in mechanically ventilated patients: a prospective observational cohort study. J Crit Care. 2013 Oct;28(5):647-54. doi: 10.1016/j.jcrc.2013.03.010. Epub 2013 May 15. PMID 23683560
- [Background] Aggarwal NR, Brower RG, Hager DN, Thompson BT, Netzer G, Shanholtz C, Lagakos A, Checkley W; National Institutes of Health Acute Respiratory Distress Syndrome Network Investigators. Oxygen Exposure Resulting in Arterial Oxygen Tensions Above the Protocol Goal Was Associated With Worse Clinical Outcomes in Acute Respiratory Distress Syndrome. Crit Care Med. 2018 Apr;46(4):517-524. doi: 10.1097/CCM.0000000000002886. PMID 29261565
- [Background] de Graaff AE, Dongelmans DA, Binnekade JM, de Jonge E. Clinicians' response to hyperoxia in ventilated patients in a Dutch ICU depends on the level of FiO2. Intensive Care Med. 2011 Jan;37(1):46-51. doi: 10.1007/s00134-010-2025-z. Epub 2010 Sep 28. PMID 20878146
- [Background] Hochberg CH, Semler MW, Brower RG. Oxygen Toxicity in Critically Ill Adults. Am J Respir Crit Care Med. 2021 Sep 15;204(6):632-641. doi: 10.1164/rccm.202102-0417CI. PMID 34086536
- [Background] Fawzy A, Wu TD, Wang K, Robinson ML, Farha J, Bradke A, Golden SH, Xu Y, Garibaldi BT. Racial and Ethnic Discrepancy in Pulse Oximetry and Delayed Identification of Treatment Eligibility Among Patients With COVID-19. JAMA Intern Med. 2022 Jul 1;182(7):730-738. doi: 10.1001/jamainternmed.2022.1906. PMID 35639368
- [Background] Wong AI, Charpignon M, Kim H, Josef C, de Hond AAH, Fojas JJ, Tabaie A, Liu X, Mireles-Cabodevila E, Carvalho L, Kamaleswaran R, Madushani RWMA, Adhikari L, Holder AL, Steyerberg EW, Buchman TG, Lough ME, Celi LA. Analysis of Discrepancies Between Pulse Oximetry and Arterial Oxygen Saturation Measurements by Race and Ethnicity and Association With Organ Dysfunction and Mortality. JAMA Netw Open. 2021 Nov 1;4(11):e2131674. doi: 10.1001/jamanetworkopen.2021.31674. PMID 34730820
- [Background] de Jonge E, Peelen L, Keijzers PJ, Joore H, de Lange D, van der Voort PH, Bosman RJ, de Waal RA, Wesselink R, de Keizer NF. Association between administered oxygen, arterial partial oxygen pressure and mortality in mechanically ventilated intensive care unit patients. Crit Care. 2008;12(6):R156. doi: 10.1186/cc7150. Epub 2008 Dec 10. PMID 19077208
- [Background] Damiani E, Adrario E, Girardis M, Romano R, Pelaia P, Singer M, Donati A. Arterial hyperoxia and mortality in critically ill patients: a systematic review and meta-analysis. Crit Care. 2014 Dec 23;18(6):711. doi: 10.1186/s13054-014-0711-x. PMID 25532567
- [Background] Mikkelsen ME, Christie JD, Lanken PN, Biester RC, Thompson BT, Bellamy SL, Localio AR, Demissie E, Hopkins RO, Angus DC. The adult respiratory distress syndrome cognitive outcomes study: long-term neuropsychological function in survivors of acute lung injury. Am J Respir Crit Care Med. 2012 Jun 15;185(12):1307-15. doi: 10.1164/rccm.201111-2025OC. Epub 2012 Apr 6. PMID 22492988
- [Background] Panwar R, Hardie M, Bellomo R, Barrot L, Eastwood GM, Young PJ, Capellier G, Harrigan PW, Bailey M; CLOSE Study Investigators; ANZICS Clinical Trials Group. Conservative versus Liberal Oxygenation Targets for Mechanically Ventilated Patients. A Pilot Multicenter Randomized Controlled Trial. Am J Respir Crit Care Med. 2016 Jan 1;193(1):43-51. doi: 10.1164/rccm.201505-1019OC. PMID 26334785
- [Background] Girardis M, Busani S, Damiani E, Donati A, Rinaldi L, Marudi A, Morelli A, Antonelli M, Singer M. Effect of Conservative vs Conventional Oxygen Therapy on Mortality Among Patients in an Intensive Care Unit: The Oxygen-ICU Randomized Clinical Trial. JAMA. 2016 Oct 18;316(15):1583-1589. doi: 10.1001/jama.2016.11993. PMID 27706466
- [Background] ICU-ROX Investigators and the Australian and New Zealand Intensive Care Society Clinical Trials Group; Mackle D, Bellomo R, Bailey M, Beasley R, Deane A, Eastwood G, Finfer S, Freebairn R, King V, Linke N, Litton E, McArthur C, McGuinness S, Panwar R, Young P; ICU-ROX Investigators the Australian and New Zealand Intensive Care Society Clinical Trials Group. Conservative Oxygen Therapy during Mechanical Ventilation in the ICU. N Engl J Med. 2020 Mar 12;382(11):989-998. doi: 10.1056/NEJMoa1903297. Epub 2019 Oct 14. PMID 31613432
- [Background] Schjorring OL, Klitgaard TL, Perner A, Wetterslev J, Lange T, Siegemund M, Backlund M, Keus F, Laake JH, Morgan M, Thormar KM, Rosborg SA, Bisgaard J, Erntgaard AES, Lynnerup AH, Pedersen RL, Crescioli E, Gielstrup TC, Behzadi MT, Poulsen LM, Estrup S, Laigaard JP, Andersen C, Mortensen CB, Brand BA, White J, Jarnvig IL, Moller MH, Quist L, Bestle MH, Schonemann-Lund M, Kamper MK, Hindborg M, Hollinger A, Gebhard CE, Zellweger N, Meyhoff CS, Hjort M, Bech LK, Grofte T, Bundgaard H, Ostergaard LHM, Thyo MA, Hildebrandt T, Uslu B, Solling CG, Moller-Nielsen N, Brochner AC, Borup M, Okkonen M, Dieperink W, Pedersen UG, Andreasen AS, Buus L, Aslam TN, Winding RR, Schefold JC, Thorup SB, Iversen SA, Engstrom J, Kjaer MN, Rasmussen BS; HOT-ICU Investigators. Lower or Higher Oxygenation Targets for Acute Hypoxemic Respiratory Failure. N Engl J Med. 2021 Apr 8;384(14):1301-1311. doi: 10.1056/NEJMoa2032510. Epub 2021 Jan 20. PMID 33471452
- [Background] Seitz KP, Wang L, Casey JD, Markus SA, Jackson KE, Qian ET, Self WH, Rice TW, Semler MW. Pulse Oximetry and Race in Critically Ill Adults. Crit Care Explor. 2022 Sep 14;4(9):e0758. doi: 10.1097/CCE.0000000000000758. eCollection 2022 Sep. PMID 36128001
- [Background] Eastwood GM, Peck L, Young H, Suzuki S, Garcia M, Bellomo R. Intensive care clinicians' opinion of conservative oxygen therapy (SpO(2) 90-92%) for mechanically ventilated patients. Aust Crit Care. 2014 Aug;27(3):120-5. doi: 10.1016/j.aucc.2013.11.004. Epub 2013 Dec 24. PMID 24369915
- [Background] Helmerhorst HJ, Schultz MJ, van der Voort PH, Bosman RJ, Juffermans NP, de Jonge E, van Westerloo DJ. Self-reported attitudes versus actual practice of oxygen therapy by ICU physicians and nurses. Ann Intensive Care. 2014 Jul 25;4:23. doi: 10.1186/s13613-014-0023-y. eCollection 2014. PMID 25512878
- [Background] Helmerhorst HJ, Schultz MJ, van der Voort PH, Bosman RJ, Juffermans NP, de Wilde RB, van den Akker-van Marle ME, van Bodegom-Vos L, de Vries M, Eslami S, de Keizer NF, Abu-Hanna A, van Westerloo DJ, de Jonge E. Effectiveness and Clinical Outcomes of a Two-Step Implementation of Conservative Oxygenation Targets in Critically Ill Patients: A Before and After Trial. Crit Care Med. 2016 Mar;44(3):554-63. doi: 10.1097/CCM.0000000000001461. PMID 26562347
- [Background] Suzuki S, Eastwood GM, Glassford NJ, Peck L, Young H, Garcia-Alvarez M, Schneider AG, Bellomo R. Conservative oxygen therapy in mechanically ventilated patients: a pilot before-and-after trial. Crit Care Med. 2014 Jun;42(6):1414-22. doi: 10.1097/CCM.0000000000000219. PMID 24561566
- [Background] Pannu SR. Too Much Oxygen: Hyperoxia and Oxygen Management in Mechanically Ventilated Patients. Semin Respir Crit Care Med. 2016 Feb;37(1):16-22. doi: 10.1055/s-0035-1570359. Epub 2016 Jan 28. PMID 26820270
- [Background] Baker DW, Persell SD. Criteria for waiver of informed consent for quality improvement research. JAMA Intern Med. 2015 Jan;175(1):142-3. doi: 10.1001/jamainternmed.2014.6977. No abstract available. PMID 25560946
- [Background] McKinney RE Jr, Beskow LM, Ford DE, Lantos JD, McCall J, Patrick-Lake B, Pletcher MJ, Rath B, Schmidt H, Weinfurt K. Use of altered informed consent in pragmatic clinical research. Clin Trials. 2015 Oct;12(5):494-502. doi: 10.1177/1740774515597688. Epub 2015 Sep 15. PMID 26374677
- [Background] Schmidt AF, Finan C. Linear regression and the normality assumption. J Clin Epidemiol. 2018 Jun;98:146-151. doi: 10.1016/j.jclinepi.2017.12.006. Epub 2017 Dec 16. PMID 29258908
- [Background] Hooper R, Teerenstra S, de Hoop E, Eldridge S. Sample size calculation for stepped wedge and other longitudinal cluster randomised trials. Stat Med. 2016 Nov 20;35(26):4718-4728. doi: 10.1002/sim.7028. Epub 2016 Jun 28. PMID 27350420